CLINICAL TRIAL: NCT07066592
Title: Investigation of the Effects of Prehabilitation Education Delivered Through a Mobile Compatible Website on Quality of Life and Symptoms in Patients Undergoing Hematopoietic Stem Cell Transplantation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Collaborators: Ankara Oncology Research and Training Hospital (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2024-11/74
Record Dates: First submitted 2025-06-25; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2024-12

CONDITIONS: Hematological Malignancy; Prehabilitation; Patient Education
Keywords: prehabilitation; quality of life; bone marrow transplantation; education
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation education provided via mobile compatible website (Experimental): Participants will receive access to the educational website containing information on the stem cell transplantation process, consisting of 9 sections, one week prior to hospital admission.
  Interventions: Behavioral: Prehabilitation education provided via mobile compatible website
- Control (No Intervention): Participants will receive routine care.

INTERVENTIONS:
Behavioral: Prehabilitation education provided via mobile compatible website — The prehabilitation education delivered through a mobile-compatible website was developed specifically for patients who are candidates for stem cell transplantation. Through this platform, patients can easily and quickly access accurate information on managing potential symptoms during the transplant process, as well as guidance on nutrition and exercise aimed at improving their quality of life.
  Arms: Prehabilitation education provided via mobile compatible website

SUMMARY:
Aim of the Study:

The aim of this study is to examine the effect of prehabilitation education delivered via a mobile-compatible website on the quality of life and symptom evaluation of patients undergoing hematopoietic stem cell transplantation (HSCT).

Research Questions:

What is the effect of prehabilitation education delivered via a mobile-compatible website on the quality of life of stem cell transplant patients? What is the effect of prehabilitation education delivered via a mobile-compatible website on the symptom management of stem cell transplant patients?

Method:

In this study, patients will be randomly assigned to one of two groups:

One group will receive prehabilitation education through a mobile-compatible website.

The other group will receive standard educational procedures.

DETAILED DESCRIPTION:
Hematopoietic Stem Cell Transplantation (HSCT) is an intensive treatment with the potential to cure hematologic malignancies and other highly morbid diseases. However, it is also associated with significant risks of morbidity and mortality. Many HSCT patients experience a variety of physical, emotional, and cognitive symptoms, particularly during the acute recovery phase following transplantation. Gastrointestinal symptoms such as nausea, vomiting, loss of appetite, mucositis, and changes in taste often emerge during the pre-transplant conditioning period and may persist for an extended period after the transplant.

Loss of strength and pain are among the most common and severe symptoms during the acute recovery phase. Other frequently encountered symptoms include anorexia, loss of muscle mass, and fatigue. During hospitalization, HSCT patients may also experience clinically significant emotional symptoms such as anxiety, depression, or adjustment disorders. These symptoms can negatively impact patients' subjective symptom burden, treatment adherence, and length of hospital stay.

Therefore, accurate assessment and management of symptoms and risks during hospitalization are essential to minimize the symptom burden in HSCT patients. Since HSCT involves high-dose chemotherapy, prolonged hospital stays, and strict isolation protocols, transplant-specific quality of life (QoL) assessment is crucial. Evaluating QoL in transplant patients can help healthcare professionals understand patients' physical, psychological, and social well-being and identify their rehabilitation needs.

Numerous symptoms caused by the disease and HSCT, as well as transplant-specific complications, significantly reduce patients' quality of life and adversely affect long-term transplant outcomes. For this reason, it is important to prepare patients adequately before undergoing HSCT. In such cases, the concept of prehabilitation is considered essential. Prehabilitation is a clinical model that introduces rehabilitation components to patients before intensive medical interventions, aiming to optimize functionality and improve tolerance to treatment.

Cancer prehabilitation is a part of the cancer rehabilitation care process. It occurs between the time of cancer diagnosis and the start of acute treatment. It includes physical and psychological assessments to establish a baseline functional level, identify impairments, and provide interventions that promote psychological health and physical improvement to reduce the incidence and/or severity of future impairments.

The aim of this study is to investigate the effect of prehabilitation education provided via a mobile-compatible website on the quality of life and symptom evaluation of patients undergoing HSCT. Patients will be randomly assigned to two groups: one group will receive prehabilitation education via a mobile-compatible website, while the other group will receive standard education procedures.

Both groups will be assessed using the Functional Assessment of Cancer Therapy-Bone Marrow Transplantation (FACT-BMT) and the Edmonton Symptom Assessment Scale (ESAS) on the day of hospital admission, the day of transplantation, and the day of discharge.

The web-based educational content consists of 9 sections:

What is stem cell transplantation? Pre-transplant preparation period Stem cell transplantation procedure and engraftment What is oral mucositis (mouth sores)? How to perform oral care? What is the risk of infection? How to protect yourself from infection? Side effects of transplant treatment Nutrition and food preparation after transplantation Returning home after stem cell transplantation and home exercise suggestions before transplant At the end of the study, the test results of the patient groups will be compared both within and between groups. The study aims to determine whether the group receiving prehabilitation education through a mobile-compatible website differs significantly from the group receiving standard education and to evaluate the impact of the educational intervention on patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing Hematopoietic Stem Cell Transplantation (HSCT) for the first time
* Having no musculoskeletal problems that would prevent physical activity
* Volunteering to participate in the study
* Between 18 and 70 years of age
* Having access to and the ability to use a mobile phone and the internet
* Literate in Turkish (able to read and write in Turkish)

Exclusion Criteria:

* Having a condition that prevents effective communication
* Being illiterate (unable to read and write)
* Inability to use technology

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2024-12-13 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
symptom management | The baseline and average 3-4 weeks
  Edmonton Symptom Assessment Scale. Each symptom is evaluated using numerical ratings ranging from 0 to 10. A score of 0 indicates that the symptom is absent, while a score of 10 indicates that the symptom is felt very severely. The severity of the symptom increases progressively from 0 to 10. (The changes will be evaluated from the baseline level to the day of transplantation and up to the day of discharge. This period takes approximately 3-4 weeks on average)
quality of functionality | The baseline and average 3-4 weeks
  Functional Assessment of Cancer Therapy-Bone Marrow Transplant (4th version) The minimum score obtainable from the FACT-BMT scale is 0, and the maximum score is 148. Higher scores indicate a better quality of life. (The changes will be evaluated from the baseline level to the day of transplantation and up to the day of discharge. This period takes approximately 3-4 weeks on average)

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Oncology Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Normann AJ, Mo CC, Wilson RL, Perez M, Cutler C, Uno H, Thompson LV, Skinner TL, Richardson PG, Marinac CR, Dieli-Conwright CM. Prehabilitation Exercise Training to Target Improved Muscle Strength in Pretransplant Patients Diagnosed With Multiple Myeloma: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2024 Dec 19;13:e64905. doi: 10.2196/64905. PMID 39701583
- [Background] Naumann K, Singh B, Bushaway S, Crane R, Deepak S, Hartland A, Konstantopoulos P, Mansell E, Marinelli V, Pallotta V, Tolfts A, Virieux A, Wall M, Wilksch S, Zhuang M, Atkinson M, Maher C. Investigating the impact of multidisciplinary prehabilitation on deconditioning in patients eligible for haematopoietic allogenic stem cell transplantation: protocol for a feasibility trial. BMJ Open. 2024 Sep 5;14(9):e084372. doi: 10.1136/bmjopen-2024-084372. PMID 39237275
- [Background] Dennett AM, Porter J, Ting SB, Taylor NF. Prehabilitation to improve function after autologous stem cell transplantation: A pilot randomized controlled trial (PIRATE). Support Care Cancer. 2025 Feb 7;33(3):164. doi: 10.1007/s00520-025-09179-1. PMID 39920425